CLINICAL TRIAL: NCT02851979
Title: PREMODEUR. "Odors to Insufflate Life". Implementation of a Controlled Olfactory Sensorial Method to Decrease Apneas in Premature Newborns. Proof of Concept Study. Latin-square Open Study With Blind Evaluation of Primary Outcome.
Brief Title: Odors to Insufflate Life
Acronym: PREMODEUR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: few inclusions - DSMB recommendation
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL16_0078
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Premature Newborns With Gestational Age 28 to 33 Weeks
Keywords: premature newborns; apneas prevention; olfactory stimulation; latin square design

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- S0 - S1 - S2 (Experimental): S0 = no stimulation; washout; S1 = vehicle; washout; S2 = olfactory stimulation
  Interventions: Other: Olfactory stimulations
- S0 - S2 - S1 (Experimental): S0 = no stimulation; washout; S2 = olfactory stimulation; washout; S1 = vehicle
  Interventions: Other: Olfactory stimulations
- S1 - S0 - S2 (Experimental): S1 = vehicle; washout; S0 = no stimulation; washout; S2 = olfactory stimulation
  Interventions: Other: Olfactory stimulations
- S1 - S2 -S0 (Experimental): S1 = vehicle; washout; S2 = olfactory stimulation; washout; S0 = no stimulation
  Interventions: Other: Olfactory stimulations
- S2 - S0 - S1 (Experimental): S2 = olfactory stimulation; washout; S0 = no stimulation; washout; S1 = vehicle
  Interventions: Other: Olfactory stimulations
- S2 - S1 - S0 (Experimental): S2 = olfactory stimulation; washout; S1 = vehicle; washout S0 = no stimulation
  Interventions: Other: Olfactory stimulations

INTERVENTIONS:
Other: Olfactory stimulations — Odors are disseminated using a portable fragrance device, a prototype developed by a research unit, CNRS UMR5292. The device is outside the incubator, the only part inside is a disposable Teflon tube. The odor flux stimulates distally the NBs' nostrils. Odoriferous compounds are placed in glass tubes. This allows the olfactometer to deliver three distinct odors (to avoid habituation) in a random scheme: spearmint odor, vanilla odor, and grapefruit odor (chemicals registered by Chemical Abstracts Service), while controlling for intensity (amount of compound), duration, and odor sequence. For the vehicle period, the glass tubes remain empty.
  Stimulations occur every 5 minutes, for 5 seconds, they are mixed in medical gas to avoid infection. There are three 24-hour periods, and two 24-hour wash out periods, followed by a maximum of 3 days of surveillance.

SUMMARY:
Apneas concern about 85% of premature newborns (NB) born after less than 34 weeks of pregnancy. They are considered as an important risk factor for subsequent neuropsychological deficiency. Current pharmacological treatments are not very effective, and have side effects (agitation, irritability, sleep disorders, tachycardia). Some studies suggest that in NBs with apneas resisting to drugs, a permanent odorisation with a drop of vanillin on the incubator's pillow might reduce the frequency of apneas. This latin square design study will test a controlled olfactory stimulation method, i.e. an olfactometer which controls the odor duration, intensity, and sequence using three different odors, to reduce apneic episodes measured using 24-registration of heart and respiratory rates.

ELIGIBILITY:
Inclusion Criteria:

* Newborns from a single or multiple pregnancy
* Newborns hospitalized in the Lyon East or Saint-Etienne neonatology services, of both sexes, born before 33 weeks of amenorrhea and after at least 6 days of life, without respiratory disease beside premature birth.
* Newborns must present at least 3 bradycardia during 3 days, or presenting apneas at observation.
* Newborns will be randomized if they present at least 3 apnea episodes per 24 hour monitored by RECAN for 3 consecutive days prior to randomization.
* Written informed consents obtained from the newborns parents or legal representatives

Exclusion Criteria:

* Severe congenital malformation
* History of allergic reaction to smell stimulation (cough, sneeze, watery eyes, breathing pauses)
* No social insurance

Min Age: 6 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Number of respiratory pauses between S1 and S2 | per 24hours
  variation of the number of apnea episodes per 24hours -registered on the continuous heart / respiratory monitoring device, defined as a total cessation of breathing superior to 20 seconds (single apnea) or ≤ 20 seconds with decreased heart rate <80 beats / min) - between olfactory stimulation (S2) and placebo stimulation (S1).

SECONDARY OUTCOMES:
difference of the number of apnea episodes between S1 and S2 | per 24hours
  difference of the number of apnea episodes between S1 and S2 adjusted on the order of stimulations, gestational age, concomitant treatments likely to interfere with breathing and their dosage
difference of the number of apnea episodes between S0 and S2 | per 24hours
  difference in the number of apnea episodes between olfactory stimulation (S2) and no stimulation (S0)
adverse events | up to day 8

CONTACTS AND LOCATIONS:
Overall Officials: HELENE GAUTHIER MOULINIER, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Hopital Femme Mère Enfant, Bron
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duchamp-Viret P, Nguyen HK, Maucort-Boulch D, Remontet L, Guyon A, Franco P, Cividjian A, Thevenet M, Iwaz J, Galletti S, Kassai B, Cornaton E, Plaisant F, Claris O, Gauthier-Moulinier H. Protocol of controlled odorant stimulation for reducing apnoeic episodes in premature newborns: a randomised open-label Latin-square study with independent evaluation of the main endpoint (PREMODEUR). BMJ Open. 2021 Sep 13;11(9):e047141. doi: 10.1136/bmjopen-2020-047141. PMID 34518252